CLINICAL TRIAL: NCT02211404
Title: Children's Sleep in the ICU
Status: Completed | Type: Observational
Sponsor: James Hungerford (Other)
Responsible Party: Sponsor-Investigator, James Hungerford, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: 13-00326
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Children Admitted to the Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Prospective evaluation of sleep in children admitted to the Intensive Care Unit at Nationwide Children's Hospital to determine how children sleep while admitted to the Intensive Care Unit

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to the Intensive Care Unit, or soon to be admitted to the ICU
* Age from 0 days to 17 years 364 days at the time of enrollment
* Any patient with anticipated ICU stay of at least overnight with a minimum of 12 hours duration

Exclusion Criteria:

* Any patient with Admitted with Traumatic Brain Injury, Admitted with an Active Seizure Disorder, Severe Developmental Delay that might impair normal sleep architecture, Known abnormal EEG, any patient actively receiving Mechanical Ventilation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | 24 Hours